CLINICAL TRIAL: NCT04423952
Title: Validity of the French Version of the Quality of Life Questionnaire COMQ12-FR
Acronym: COMQ12-FR
Status: Withdrawn | Type: Observational
Why Stopped: The study never started
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200195; 2019-A00377-50 (Other: ID RCB (ANSM))
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-10

CONDITIONS: Chronic Otitis Media
Keywords: Chronic otitis media in children; Standardized quality of life measurement questionnaire
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with chronic otitis media: Patients aged 7 to 15 years with chronic otitis media.
  Interventions: Other: COMQ-12 questionnaire
- Controls: Minors aged 7 to 15 years, with no and no history of chronic otitis.
  Interventions: Other: COMQ-12 questionnaire

INTERVENTIONS:
Other: COMQ-12 questionnaire — Subjects respond to COMQ-12 questionnaire twice at 15 days apart. COMQ-12 : quality of life measurement questionnaire related to chronic otitis media.
  Other Names: Patient questionnaire

SUMMARY:
The World Health Organization estimates that chronic otitis media could reach between 65 and 350 million people worldwide and thus be an important cause of medical consultation and prescription drugs.

The medical care of chronic otitis is difficult, despite several medical and surgical treatment options. Moreover this pathology is gladly recurrent.

The completion of a standardized questionnaire to track symptoms objectively over time is fundamental to verify the efficacy of specific treatments and to compare treatments.

The quality of life measurement questionnaire related to chronic otitis media (COMQ-12) is a new questionnaire, validated in English, to assist the physician in evaluating chronic otitis media.

The objective of this study is to translate and validate the test in French in children.

DETAILED DESCRIPTION:
The World Health Organization estimates that chronic otitis media could reach between 65 and 350 million people worldwide and thus be an important cause of medical consultation and prescription drugs.

The medical care of chronic otitis is difficult, despite several medical and surgical treatment options. Moreover this pathology is often recurrent.

The completion of a standardized questionnaire to track symptoms objectively over time is fundamental to verify the efficacy of specific treatments and to compare treatments.

The quality of life measurement questionnaire related to chronic otitis media (COMQ-12) is a new questionnaire, validated in English, to assist the physician in evaluating chronic otitis media.

The original version of the COMQ12 questionnaire, in English, was developed by Phillips et al.. The construction of this questionnaire was based on three other questionnaires : the Chronic Ear Survey (CES), the Chronic Otitis Media Outcome-15 (COMOT-15), and the Chronic Otitis Media-5 (COM-5). The initial validation of the English version of Phillips et al. was evaluated with an alpha value of Cronbach to 0.889, which shows high internal consistency and would allow its use in several reputed international centers of otology.

The objective of this study is to translate and validate the test in French in children.

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 7 to 15 years (inclusive)
* Patients with chronic otitis media, united or bilateral
* Controls: subjects without chronic otitis media or any other pathology of the ear at the time of Inclusion or in background
* holders of parental authority not opposed to participation in the study

Exclusion Criteria:

- Non-comprehension of french

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the department of otolaryngology and cervico-facial surgery of Necker-Enfants Malades hospital and siblings for the control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Reproducibility | 1 year
  Reproducibility of the questionnaire completed by a subject at 15 days apart. Student t-test. COMQ12 : Chronic Otitis Media Questionnaire 12. Score range from 0 to 110 (0 is the score in the absence of symptoms, 110 the worst possible).
Consistency reliability test | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
  COMQ12 : Chronic Otitis Media Questionnaire 12. Score range from 0 to 110 (0 is the score in the absence of symptoms, 110 the worst possible).
Item-total Pearson correlation | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
  COMQ12 : Chronic Otitis Media Questionnaire 12. Score range from 0 to 110 (0 is the score in the absence of symptoms, 110 the worst possible).
Principal components analysis | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
  COMQ12 : Chronic Otitis Media Questionnaire 12. Score range from 0 to 110 (0 is the score in the absence of symptoms, 110 the worst possible).

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Denoyelle, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No